CLINICAL TRIAL: NCT06177509
Title: Effect of Graded Aerobic Exercise in Mild Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Oslo University Hospital (Other); Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gradert trening ved mTBI
Record Dates: First submitted 2023-12-05; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury
Keywords: post-concussion symptoms; autonomic nervous system dysfunction; Buffalo concussion treadmill test
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind parallel group design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group - Graded Aerobic Exercise (Experimental): Participants will follow a sub-symptom aerobic exercise program (approx. 30 min) 3 - 5 times pr week for twelve weeks. Sub-symptom threshold aerobic exercise means to exercise at 80-90% of the maximum threshold heart rate achieved during the BCTT. To ensure proper exercise dose and progression, participants will be retested every three weeks. During the first three weeks, the participants will be offered one weekly guided exercise session. The other 2 - 4 weekly sessions the participants will carry out on their own, choosing activities based on experience, preferences and possibilities (e.g. walking, jogging, stationary bike, swimming). The intensity of the sub-symptom threshold aerobic exercise will be monitored using a heart rate monitor and the BORG scale. Compliance with the sub-symptom threshold aerobic exercise program will be recorded by the patients in an exercise diary, which is followed up by a weekly reminder over the phone/sms by a physiotherapist in the project.
  Interventions: Other: Graded Aerobic Exercise
- Control group - Outpatient multidisciplinary follow-up (Treatment as usual - TAU) (No Intervention): TAU includes assessment and treatment provided by a multidisciplinary outpatient rehabilitation team. Patients will undergo a medical examination and assessment of physical, cognitive, and mental health and functioning, followed by individually adapted rehabilitation program. The interdisciplinary team consists of a specialist in physical medicine and rehabilitation, (neuro)psychologist, occupational therapist, physiotherapist, and social worker. The main focus is on improving the level of function in everyday life and gradual return to work and education.

INTERVENTIONS:
Other: Graded Aerobic Exercise — Participants will follow a sub-symptom aerobic exercise program (approx. 30 min) 3 - 5 times pr week for twelve weeks. Sub-symptom threshold aerobic exercise means to exercise at 80-90% of the maximum threshold heart rate achieved during the BCTT. To ensure proper exercise dose and progression, participants will be retested every three weeks. During the first three weeks, the participants will be offered one weekly guided exercise session. The other 2 - 4 weekly sessions the participants will carry out on their own, choosing activities based on experience, preferences and possibilities (e.g. walking, jogging, stationary bike, swimming). The intensity of the sub-symptom threshold aerobic exercise will be monitored using a heart rate monitor and the BORG scale. Compliance with the sub-symptom threshold aerobic exercise program will be recorded by the patients in an exercise diary, which is followed up by a weekly reminder over the phone/sms by a physiotherapist in the project.
  Arms: Intervention group - Graded Aerobic Exercise

SUMMARY:
There is a paucity of knowledge about mechanisms behind mild traumatic brain injury (mTBI) subgroup's sustained problems, and effective interventions that can alleviate this disabling condition. Persistent Post-concussive Symptoms (PCS) affect between 20% and 30% of individuals after mTBI.

This Randomized Controlled Trial (RCT) will investigate whether graded aerobic exercise has a positive effect on symptom burden (including exercise intolerance) and Autonomic Nervous System (ANS) dysfunction in patients with PCS.

This study will expand upon previous work on adolescents with sport-related concussion in the acute phase. It will cover a wider age group and will include patients with persisting symptoms, thus providing knowledge on whether a sub-symptom threshold aerobic exercise program will alleviate symptom burden in adult patients with PCS.

Furthermore - looking into the relationship between mTBI and ANS function, this study is expected to contribute to a better understanding of the neurobiological factors involved in PCS. The results may also help developing targeted interventions to specific characteristics in persistent symptoms after mTBI.

DETAILED DESCRIPTION:
Background: TBI is a public health challenge of considerable, but insufficiently recognized proportions. Therefore, a concerted effort should be made to reduce the burden and impact of TBI. Health care providers are in need of standardization of the medical examination and targeted individual interventions with potential to treat PCS.

Main purpose: The main purpose of this study is to evaluate whether a progressive, sub-symptom threshold aerobic exercise program in addition to ordinary rehabilitation will lead to clinically meaningful reduction in symptom burden, normalize exercise tolerance and improve health-related quality of life compared to a control group that only receives ordinary rehabilitation. In addition, changes in ANS function will be assessed in both the intervention and the control group.

Design: Randomized, controlled, single-blind parallel-group study with two measurement points; T0 at baseline and T1 after the intervention.

Method: The Buffalo Concussion Treadmill Test (BCTT) will be used to expose exercise intolerance, and participants with exercise intolerance will be randomized to the intervention group or the control group. Both groups will receive ordinary rehabilitation. The intervention group will in addition receive an individualized (based on BCTT) sub-symptom threshold aerobic exercise program for 12 weeks. To assess ANS function, Arterial spin labeling (ASL) MRI and Cold Pressor Test (CPT) will be performed at T0 and T1. Symptom burden will be assessed by Rivermead Post-concussion Symptom Questionnaire (RPQ) and other patient reported outcomes measurements including self-reported autonomic symptoms (the Composite Autonomic Symptom Score 31) will also be used.

Clinical relevance: Self-reported ANS, exercise intolerance testing, the CPT and ASL-MRI could prove to be useful clinical assessment tools to confirm the PCS-diagnosis and to determine readiness to return to preinjury level of day-to-day activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild TBI as defined by the World Health Organization (WHO)
* Diagnosis of PCS based on ICD-10 criteria for a minimum of 3 months to a maximum of 2 years
* Age 18-60 years.
* Reduced tolerance to physical activity/exercise intolerance (self-reported worsening of symptoms such as dizziness, nausea or headache during physical activity and exercise). Or have not yet tried physical activity/exercise after the injury.

Exclusion Criteria:

* Other neurological or severe psychiatric conditions listed in the medical record.
* Heart-lung disease.
* Extremity injuries that prevent physical exercise
* Drug addiction
* Insufficient understanding of the Norwegian language (unable to follow instructions and/or fill in forms).
* Normal BCTT.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change on the Rivermead Post-concussion Symptom Questionnaire (RPQ) | Baseline and 12 weeks
  A 16-item standardized and validated questionnaire designed to measure the severity of post-concussive symptoms following mTBI. The five-point ordinal scale ranges from 0 (no problem) to 4 (severe problem). The total score ranges from 0-64, with higher scores indicating a higher symptom load. RPQ has satisfactory psychometric properties and is widely used in mTBI and persistent post-concussive symptoms research. The minimal clinically important difference (MCID) is 4,6 points.

SECONDARY OUTCOMES:
Change on the Cold Pressor Test Cold Pressor Test | Baseline and 12 weeks
  The CPT is a test of ANS sympathetic activation that has been used to study a variety of populations. Submerging the hand in cold water stimulates the cold-sensitive nociceptive fibres, resulting in increased sympathetic neural activity, which will raise heart rate and blood pressure. Blunted and delayed cardiovascular responses, when compared to healthy subjects data, indicates ANS dysfunction. The participant's hand is submerged in ice water (approx. 0°C) for 120 seconds. Prior to, during, and after cooling of the hand, beat-to-beat blood pressure is measured by finger photoplethysmography (Finapres® NOVA; Finapres Medical Systems BV, Netherlands) and a three-lead electrocardiography (model DA100C; Biopac Systems Inc, Goleta, CA) is used to continuously record heart rate.
Change on Arterial spin labeling (ASL) | Baseline and 12 weeks
  ASL MRI is an MRI sequence to quantitatively assess CBF. Alterations in CBF is well documented in moderate/severe TBI, and has been identified in animal models of mTBI and in children and athletes in the acute/subacute phase after mTBI. ANS sympathetic activation constricts and parasympathetic activation dilates cerebral blood vessels in turn altering CBF, which can be revealed by ASL. The scans will be performed on a 3.0T MRI scanner (Signa HDx, GE Medical Systems, Milwaukee, Wisconsin). The 3D ASL scan will automatically be processed into quantitative maps of global and regional CBF. Due to restricted resources, approximately 1/3 of the participants in each group (10 - 15 pr group) will be randomly allocated to an ASL MRI assessment at T0 and T1.
Change on the Buffalo Concussion Treadmill Test (BCTT) | Baseline and 12 weeks
  The BCTT is a standardized incremental test of exercise tolerance. Exercise tolerance is tested by gradually increasing the load while walking on a treadmill. The test starts with speed set at 5.2 or 5.8 km/h (determined by participant's height) at 0% incline for the first minute. The speed is maintained and the incline is increased by 1% each minute. Every minute, overall post-concussion symptom burden is registered using a 0-10 numeric rating scale (NRS), rating of perceived exertion is obtained using Borg Rating of Perceived Exertion (RPE) and heart rate (HR) is obtained using a PolarH10 HR monitor. The test is stopped at symptom exacerbation defined as an increase of ≥ 3 points on the NRS (positive test). If voluntary exhaustion (RPE ≥ 17 on the 6 - 20 Borg rating scale) or 90% of age predicted maximum HR is reached without symptom exacerbation the test is stopped (negative test).Outcome measures from the BCTT are HR at- and time until stopping criteria are reached.
Change on 0-10 Numeric Rating Scale (NRS) in Concussion Symptom Burden | Baseline and 12 weeks
  Reported concussion-specific symptoms during incremental tredmill test (BCTT) on a scale from 0 - 10, where 0 means no symptoms and 10 means worst symptoms ever experienced.
Change on Borg scale - Rating of Perceived Exertion (RPE) | Baseline and 12 weeks
  Reported Percived Exortion during incremental tredmill test (BCTT) on a scale from 6- 20, 6 being no exertion and 20 being the maximum exortion.
Change in Heartrate (HR) | Baseline and 12 weeks
  Heartrate is obtained by a Polar OH chest band HR monitor during incremental tredmill test (BCTT).

OTHER OUTCOMES:
Change on the Composite Autonomic Symptom Score 31 (COMPASS 31) | Baseline and 12 weeks
  This is a 31-item self-assessment questionnaire assessing autonomic symptoms in six domains, orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder, and pupillomotor function. The sum of the six weighted sub-scores yields the total weighted score from 0 to 100, with 0 meaning no autonomic symptoms, and 100 reflecting the most severe autonomic symptoms.
Change on the Quality of life after TBI (Qolibri) OA scale | Baseline and 12 weeks
  Assesses overall satisfaction with facets of life relevant to persons with TBI. The six-item questionnaire covers physical condition, cognition, emotions, function in daily life, personal and social life, current situation and future prospects. Each item is scored from 1 (not at all) to 5 (very). The sum is converted arithmetically to a percentage scale from 0-100 (worst-best) .
Change on the International Physical Activity Questionnaires (IPAQ) | Baseline and 12 weeks
  Will be used to obtain data on health-related physical activity. It contains 4 items regarding time spent on vigorous activities, moderate activities, walking and sitting during the last 7 days.
Change on the Patient Health Questionnaire (PHQ-9) | Baseline and 12 weeks
  Assesses symptoms of depression. The tool contains 9 items, has a scale range from 0 to 27, and has been validated. It is commonly used in individuals with mild to severe TBI.
Change on the Generalized Anxiety Disorder Scale (GAD-7) | Baseline and 12 weeks
  Measures anxiety and contains 7 items and is a commonly used in the mTBI population. Scale range from 0 to 21.
Change on the Fatigue Severity Scale (FSS) | Baseline and 12 weeks
  A commonly used tool for brief assessment of fatigue interference with a scale range from 9 to 63.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Løvstad, Professor, Principal Investigator — Head of psychology
Locations (2):
- Norway (2):
  - Sunnaas rehabilitation hospital, Nesoddtangen
  - Oslo University Hospital, Oslo